CLINICAL TRIAL: NCT02938481
Title: International Prospective Observational Cohort Study for Optimal Bowel Resection Extent and Central Radicality for Colon Cancer
Acronym: T-REX
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Tokyo Medical and Dental University, Japan (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRICC1410
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer
Keywords: colon cancer, lymph node, extent of bowel resection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Resected surgical specimens to take photographs
  * Lymph nodes retrieved from Resected surgical specimens to categorise
Oversight: Data Monitoring Committee: No

SUMMARY:
The T-REX study aims to clarify the actual status of metastatic lymph node (LN) distribution in colon cancer and provide reliable evidence regarding the optimal length of bowel resection and the extent of central lymph node dissection in colon cancer surgery.

DETAILED DESCRIPTION:
In colon canser, the incidence of metastasis in the pericolic lymph nodes (LNs) located along the bowel and marginal artery is high. The optimal extent of bowel resection is closely associated with how we define 'regional' pericolic LNs, which should be resected because of the risk of metastasis. However, there are no standardised criteria for 'regional' LNs in the pericolic area.

To establish a consensus for the extent of bowel resection and appropriate central LN dissection, international prospective stdies focusing on the distribution of metastatic LNs along the bowel and the primary feeding artery are conducted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colon adenocarcinoma
* Pathological stage Ⅰ, Ⅱ or Ⅲ
* Potentially curative surgery
* Informed consent for observational data collection

Exclusion Criteria:

* Tis (mucosal cancer)
* Multiple colon cancers
* All patients with preoperative adjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colon cancer who will receive potentially curative surgery at participating institutions between 22 Jan 2015 and 22 Jan 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3647 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Distribution of metastatic LNs | At the time of patient registry in
Distribution of metastatic LNs | At the time of 4 years after surgery

SECONDARY OUTCOMES:
Prognostic outcomes according to the length of bowel resection | 4 years
Prognostic outcomes according to the central radicality | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, M.D., Ph.D, Study Director — Tokyo Medical and Dental University, Japan
Locations (36):
- University Hospital Erlangen, Erlangen, Bavaria, Germany
- Japan (27):
  - Aichi Cancer Centre Hospital, Nagoya, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - National Canser Centre Hospital East, Chiba, Chiba
  - Teikyo University Chiba Medical Center, Ichihara-shi, Chiba
  - Keiyukai Sapporo Hospital, Sapporo, Hokkaido
  - Kurume University School of Medicine, Kurume, Hukuoka-prefecture
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Saisei-kai Yokohama-shi Nanbu Hospital, Yokohama, Kanagawa
  - Yokohama-city University, Yokohama, Kanagawa
  - Kanagawa Cancer Centre Hospital, Yokohama, Kanagawa
  - Takano Hospital, Kumamoto, Kumamoto
  - Mie University Graduate School of Medicine, Tsu, Mie-ken
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka International Cancer Institute, Osaka, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - National Defense Medical College, Tokorozawa, Saitama
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Shizuoka Cancer Centre Hospital, Sunto-gun, Shizuoka
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Disease Centre Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Centre Central Hospital, Chuo-ku, Tokyo
  - Teikyo University School of Medicine, Itabashi-ku, Tokyo
  - Kyorin University School of Medicine, Mitaka, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo
  - Wakayama Medical University, Wakayama, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata
- Lithuania (2):
  - Klaipeda University hospital, Klaipėda, Lietuva
  - National Cancer Institute, Lithuania, Vilnius
- I.M. Sechenov First Moscow State Medical University, Moscow, Russia
- South Korea (2):
  - Yonsei University, Seodaemun-gu, Seoul
  - University of Ulsan College of Medicine and Asan Medical Center, Songpa-Gu, Seoul
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shiozawa M, Ueno H, Shiomi A, Kim NK, Kim JC, Tsarkov P, Grutzmann R, Dulskas A, Liang JT, Samalavicius N, West N, Sugihara K. Study protocol for an International Prospective Observational Cohort Study for Optimal Bowel Resection Extent and Central Radicality for Colon Cancer (T-REX study). Jpn J Clin Oncol. 2021 Jan 1;51(1):145-155. doi: 10.1093/jjco/hyaa115. PMID 33215206